CLINICAL TRIAL: NCT02565121
Title: Olfaction Disorders in Patients Included in The Trauma Brain Injury (TBI) Database at Trondheim University Hospital: Prevalence and Treatment
Brief Title: Olfaction Disorders in Patients Included in The Trauma Brain Injury (TBI) Database at Trondheim University Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/427
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Brain Injuries; Olfaction Disorders
Keywords: Olfactory perception; Adrenal cortex hormones; Steroids; Education
MeSH Terms: conditions — Brain Injuries; Olfaction Disorders; Anosmia | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olfactory disorder after brain trauma (Experimental): Recruited from 250 patients with moderate to severe traumatic brain injury in the Hodeskadeprosjektet (TBI) cohort. Treatment with (first) corticosteroids and (second) olfactory stimulation.
  Interventions: Drug: corticosteroids; Behavioral: olfactory stimulation

INTERVENTIONS:
Drug: corticosteroids
Behavioral: olfactory stimulation — stimulation with odorants by sniffing 4 different odorants for a total of 5 minutes twice a day during 3 months

SUMMARY:
The aim of the study is to see whether patients with chronic smell impairment after brain injury benefit from a treatment that consists of corticosteroids, and then olfactory training in 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the TBI Database
* 18-65 years of age per 01.10. 2012
* Olfaction score by Sniffin Sticks Threshold-Discrimination-Identification (TDI) < 30 confirming dysosmia

Exclusion Criteria:

* Unable to express senses.
* Unable to follow treatment and protocol
* pregnancy
* diabetes
* tendency to infections
* hypertonia
* dyspepsia
* interfering medication (hormonal treatment, NSAIDS, antidiabetics, barbiturates, fenitoin, carbamazepin, rifampicin, cyclophosphamides)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
number of patients who have improved olfaction perception (by at least 5 points on the Threshold-Discrimination-Identification (TDI) score | 1 year
  TDI score measured by Sniffin Sticks

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kvermo, Study Director — St. Olavs Hospital
Locations (1):
- ENT department St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Bratt M, Skandsen T, Hummel T, Moen KG, Vik A, Nordgard S, Helvik AS. Frequency and prognostic factors of olfactory dysfunction after traumatic brain injury. Brain Inj. 2018;32(8):1021-1027. doi: 10.1080/02699052.2018.1469043. Epub 2018 May 9. PMID 29741969
- [Result] Bratt M, Moen KG, Nordgard S, Helvik AS, Skandsen T. Treatment of posttraumatic olfactory dysfunction with corticosteroids and olfactory training. Acta Otolaryngol. 2020 Sep;140(9):761-767. doi: 10.1080/00016489.2020.1767301. Epub 2020 Jun 3. PMID 32491937